CLINICAL TRIAL: NCT01436279
Title: Mifepristone Versus Osmotic Dilator Insertion for Cervical Preparation Prior to Surgical Abortion at 15-18 Weeks
Acronym: SaMi2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-31032; AU 6003109 (Other Grant/Funding Number: Society of Family Planning)
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Cervical Preparation
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mifepristone + misoprostol (Experimental): Mifepristone 200 mg PO given 20-24 hours prior to procedure, misoprostol 400 mcg given 2 hours prior to procedure
  Interventions: Drug: Mifepristone
- Osmotic dilators (Active Comparator): Placed 20-24 hours prior to procedure
  Interventions: Device: osmotic dilators

INTERVENTIONS:
Drug: Mifepristone — 200 mg po 20-24 hours prior to the procedure
  Other Names: Mifeprex; RU-486; Mifegyne
  Arms: Mifepristone + misoprostol
Device: osmotic dilators — osmotic dilators placed in the cervix 20-24 hours prior to the procedure
  Other Names: Laminaria; Dilapan-S; Dilapan
  Arms: Osmotic dilators

SUMMARY:
In this study the investigators plan to compare mifepristone and misoprostol use to osmotic dilator use for cervical preparation for 15-18 week surgical abortion. Mifepristone would be given 24 hours prior to abortion, and misoprostol 400 mcg would be administered buccally 2 hours prior to abortion. Osmotic dilators are the method currently used in our institution, and are placed 24 hours prior to abortion. The primary outcome will be the length of the procedure. Secondary outcomes will include amount of dilation achieved, ease of procedure, participant's assessment of discomfort before mifepristone or dilators, discomfort during the abortion procedure, acceptability to participants, and acceptability to staff.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-50 years of age undergoing surgical termination of pregnancy
* English or Spanish speaking
* Gestational age between 15 and 18 weeks gestation on day of abortion (inclusive), by ultrasound dating
* Eligible for a dilation and evacuation abortion with local anesthesia and sedation
* Ultrasound for dating purposes done within the last two weeks

Exclusion Criteria:

* Intrauterine infection
* Fetal demise
* Ruptured membranes
* Multiple gestation
* Uterine anomaly or significant distortion of the uterus with fibroids
* BMI greater than 45
* Inability to place osmotic dilators
* Active substance abuse or intoxication
* Adrenal failure, chronic corticosteroid use, anticoagulant usage
* Severe cervicitis, until treated and resolved
* Prior Cesarean section

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarita Sonalkar, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
Started | 30 | 20
Completed | 30 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators | Total
Number analyzed (Participants) | 30 | 20 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 20 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 20 | 50
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Length of Procedure
Description: Interval from speculum insertion to speculum removal
Time Frame: Subjects will be followed from the administration of mifepristone/misoprostol or laminaria, until the end of their procedure, a total of two days.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
Number analyzed (Participants) | 30 | 20
minutes | 14 [12 to 17] | 13.5 [11 to 16]

2. Secondary Outcome: Operative Time
Description: Interval from initiation of vacuum aspiration to speculum removal
Time Frame: Subjects will be followed from the administration of mifepristone/misoprostol, or laminaria, until the end of their procedure, a total of two days.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
Number analyzed (Participants) | 30 | 20
minutes | 9 [7 to 12] | 8.5 [7 to 9.5]

3. Secondary Outcome: Subject Discomfort Before the Abortion
Description: Pain was subjectively described by the subjects as : None, Mild, Moderate, Severe
Time Frame: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
Number analyzed (Participants) | 30 | 20
participants
  None | 18 | 7
  Mild | 7 | 6
  Moderate | 5 | 3
  Severe | 0 | 4

4. Secondary Outcome: Pain Medication (Fentanyl) During the Abortion
Description: Amount of pain medication used during the procedure: reported as micrograms of fentanyl
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
Number analyzed (Participants) | 30 | 20
mcg | 3.1 (1.34) | 2.9 (1)

5. Secondary Outcome: Pain Medication (Midazolam) During the Abortion
Description: Amount of pain medication used during the procedure: reported as milligrams of midazolam
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
Number analyzed (Participants) | 30 | 20
mg | 104 (31) | 105 (26)

6. Secondary Outcome: Cervical Dilation Achieved
Description: Cervical dilation at start of procedure
Time Frame: At time of abortion
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
Number analyzed (Participants) | 30 | 20
mm | 42 (11) | 56 (5)

7. Secondary Outcome: Acceptability to Patient
Description: Patient was asked whether they would choose to be in the same group again if they had a similar procedure again. The number of participants whose response was "yes" is being reported.
Time Frame: After procedure completion
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
Number analyzed (Participants) | 30 | 20
Participants | 26 | 11

8. Secondary Outcome: Difficulty of Procedure
Description: Outcome measure is the number and percentage of participants where the provider rated the procedure as "difficult or very difficult". Provider assessment of difficulty of procedure categories were: "very easy", "easy", "moderate", "difficult", or "very difficult."
Time Frame: After completion of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
Number analyzed (Participants) | 30 | 20
Participants | 5 | 3

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Mifepristone + Misoprostol | Osmotic Dilators
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/20
Other Adverse Events (participants affected / at risk) | 0/30 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes